CLINICAL TRIAL: NCT00850655
Title: Genetic Association Mapping of Malaria Resistance in Anopheles Gambiae
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0607M88827
Record Dates: First submitted 2008-10-16; First posted 2009-02-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study of the genetics of malaria transmission by the mosquito vector in Africa, Anopheles gambiae. The study focuses on the mosquito vector, not the human subjects infected with malaria. DNA extracted from infected mosquitoes will be analyzed genetically by microsatellite and single-nucleotide polymorphisms (SNPs) to identify mosquito genes that control mosquito resistance to malaria parasites.

DETAILED DESCRIPTION:
A standard diagnostic blood smear from a drop of blood will be carried out on 20 study subjects once per month. One malaria-positive subject from among the 20 will be asked to donate 5cc of blood, also no more frequently than once per month. The blood will be placed in a water-jacketed heated membrane feeding device that will be positioned on top of a cage of mosquitoes. The mosquitoes are attracted to the warmth and drink the blood through the artificial skin-like membrane. The goal of the research is to study the infected mosquitoes. No studies will be carried out on the human subjects. The point of human subjects involvement is to obtain the naturally malaria-infected blood for feeding of mosquitoes. After blood feeding, the mosquitoes are held in an environmental chamber for one week, at which time they are dissected to count numbers of malaria parasites developing on the mosquito stomach wall. This number constitutes the quantitative phenotype, and we extract genomic DNA from the carcass for genetic marker typing, which constitutes the genotype. Genetic linkage analysis identifies markers near genes that control parasite number, thus resistance or susceptibility to parasite infection.

ELIGIBILITY:
Inclusion Criteria:

* 5-10 years old, and general good health

Exclusion Criteria:

* Outside age group
* Specific diagnosable health problems
* General poor health

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
mosquito infection | one week
  Protocol involves non-invasive blood draw from participant screened by finger-prick for infection with malaria. Drawn blood (0.5cc) is placed in artificial membrane feeder for feeding of mosquitoes. Primary outcome is infection of mosquitoes, detectable one week after blood feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Vernick, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No